CLINICAL TRIAL: NCT04248283
Title: A Clinical Investigation of the Adjustable Continence Therapy (ACT) for Female Stress Urinary Incontinence Due to Intrinsic Sphincter Deficiency
Brief Title: Adjustable Continence Therapy (ACT) for the Treatment of Female SUI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uromedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UM08
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Urinary Incontinence; Urinary Incontinence,Stress
Keywords: Urinary Incontinence; Urination Disorders; Urination Involuntary; Urologic Diseases; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urination Disorders; Nocturnal Enuresis; Urologic Diseases; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: A prospective, single arm, non-randomized, multicenter, prospective case-series trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Adjustable Continence Therapy for Women (Experimental): Implantation of the Adjustable Continence Therapy for the treatment of female SUI.
  Interventions: Device: Adjustable Continence Therapy for Women (ACT)

INTERVENTIONS:
Device: Adjustable Continence Therapy for Women (ACT) — Two ACT devices are implanted in each patient. The devices are intended for implantation in the paraurethral space, with the balloons located on each side of the urethra near the bladder neck. The ports are placed subcutaneously in the labia majora. The balloons are filled after implantation with an isotonic solution via needle injection into the port. The ACT implant can be placed using local, spinal or general anesthesia with the surgical instruments (provided separately).

SUMMARY:
A prospective, single arm, non-randomized, multicenter, prospective case-series trial. The purpose of this trial is to demonstrate the safety and effectiveness of using the Adjustable Continence Therapy (ACT) to provide a clinically relevant improvement in stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Female at least 22 years old
2. Diagnosed with stress urinary incontinence with primary Intrinsic Sphincter Deficiency
3. Provocative pad weight of greater than 11.0 grams
4. Candidate for surgical intervention
5. Negative urinalysis
6. Normal cystourethroscopy
7. Failed at least 6 months of previous treatment(s) for stress urinary incontinence (e.g., exercise regimen, electrical stimulation, surgical procedures, etc). Note: patients may have failed prior anti-incontinence procedures for SUI (e.g., suspension, sling, or urethral bulking agent)
8. Willing and able to sign informed consent and comply with trial follow-up requirements

Exclusion Criteria:

1. Pregnant or lactating
2. Life expectancy of less than 5 years
3. Has uncontrolled diabetes as evidenced by HbA1c over 6.5% and fasting plasma glucose over 130 mg/dL
4. Has auto-immune disease
5. Undergoing radiation therapy
6. Active urinary tract infection
7. Detrusor instability refractory to medication
8. Reduced bladder compliance as defined by a cystometrogram
9. Significant residual volume (greater than 100 ml) after voiding in which detrusor contraction is weak, when the bladder volume is greater than or equal to 250 ml
10. Has, had, or is suspected of having bladder cancer
11. History of bladder stones
12. Urethral stricture evidenced during cystourethroscopy
13. Has a neurogenic bladder that is atonic or has detrusor sphincter dyssynergia
14. Has a diathesis, hemophilia, or a bleeding disorder
15. Has a rectocele, cystocele, urethrocele, enterocele, or pelvic prolapse of grade 3 or higher
16. Had prior pelvic radiotherapy
17. Had a prior artificial urinary sphincter implanted
18. Has a neurogenic condition known to affect bladder/sphincter function

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Provocative pad weight | 12 months
  Change in provocative pad weight from baseline

SECONDARY OUTCOMES:
Urogenital Distress Inventory (UDI) | 12 months
  Six item questionnaire. Scores range from 0-100. 0 being not distressed, 100 being very distressed.
Incontinence Quality of Life Questionnaire (I-QOL) | 12 months
  Twenty-two item questionnaire. Scores range from 0-100. 0 being lowest quality of life, 100 being highest quality of life.

OTHER OUTCOMES:
Complete adverse event profile | 12 months
  Collection of patient safety information

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C Cook, PhD, Study Director — Uromedica, Inc.
Locations (2):
- United States (2):
  - University of Colorado, Denver, Colorado
  - CHI Health Research Center, Omaha, Nebraska